CLINICAL TRIAL: NCT02745561
Title: A Phase II Study of Endostatin in Combination With Oxaliplatin and Radiotherapy in Esophageal Cancer Patients.
Brief Title: Endostatin in Combination With Oxaliplatin and Radiotherapy in Esophageal Cancer Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shixiu Wu, MD, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH05
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Cancer; Endostatin
Keywords: Endostatin; Oxaliplatin; Esophageal Cancer; chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endostatins; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoradiotherapy Arm (Experimental): Radiotherapy will be delivered with a daily fraction of 2.0 Gy to a total dose of 60 Gy over 6 weeks. Endostatin will be administered at a dose of 7.5 mg/m2/day concurrent with radiotherapy. Oxaliplatin (135mg/m², d1) will be administered on Day 1 and Day 29 of radiotherapy.
  Interventions: Drug: Endostatins; Drug: Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Endostatins — Endostatin will be administered at a dose of 7.5 mg/m2/day concurrent with radiotherapy.
Drug: Oxaliplatin — Oxaliplatin (135mg/m², d1) will be administered on Day 1 and Day 29 of radiotherapy.
Radiation: Radiotherapy — Radiotherapy will be delivered with a daily fraction of 2.0 Gy to a total dose of 60 Gy over 6 weeks.

SUMMARY:
Endostatin inhibits the pro-angiogenic action of basic fibroblast growth factor and vascular endothelial growth factor in esophageal cancer.This study aims at assessing the efficacy and safety of endostatin combined with concurrent chemoradiotherapy with Oxaliplatin in esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed esophageal carcinoma
2. Age of 18 -80
3. ECOG performance status: 0-1;
4. No treatments prior to enrollment;
5. At least one measurable lesion on CT, MRI or esophageal barium exam;
6. Normal functions of heart, lung, liver, kidney and bone marrow Blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL
7. Informed consent signed

Exclusion Criteria:

1. Prior treatments of chemotherapy or irradiation;
2. Poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable;
3. Contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis;
4. Participating in other clinical trials;
5. Pregnancy, breast feeding, or not adopting birth control;
6. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities
7. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
response rate | week 3-4
  Response rate will be done after 3-4 weeks following the last radiotherapy session.

SECONDARY OUTCOMES:
Acute and late toxicities assessed based on the common toxicity criteria for adverse events version 3.0 (CTCAEv3.0) | year 0 - year 3
  Acute and late toxicities will be assessed based on the common toxicity criteria for adverse events version 3.0 (CTCAEv3.0).
Progression-free survival | year 0 - year 3
  Progression-free survival (PFS) will be calculated from the date of chemoradiotherapy initiation to the date of documented failure (local recurrence or metastasis occurrence) or the date of the last follow-up for those remaining.
Overall survival | year 0 - year 3
  Overall survival (OS) will be determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li W, Chen P, Zhang N, Song T, Wu S. Endostatin and Oxaliplatin-Based Chemoradiotherapy for Inoperable Esophageal Squamous Cell Carcinoma: Results of a Phase II Study. Oncologist. 2019 Apr;24(4):461-e136. doi: 10.1634/theoncologist.2019-0119. Epub 2019 Mar 8. PMID 30850562